CLINICAL TRIAL: NCT03628235
Title: Indirect and Out-of-Pocket Costs of Huntington's Disease in the United States
Brief Title: HD-Charge: Indirect and Out-of-Pocket Costs of Huntington's Disease in the United States
Status: Completed | Type: Observational
Sponsor: CHDI Foundation, Inc. (Other)
Collaborators: IQVIA Company (Unknown)
Responsible Party: Sponsor
Other Study IDs: C-001117-1
Record Dates: First submitted 2018-05-29; First posted 2018-08-14 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Huntington's Disease
Keywords: online survey; indirect costs; out-of-pocket costs; HD; Huntington's disease; companions; Enroll-HD
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Early stage HDGECs: CAG length ≥ 40; DCL = 4, TFC ≥ 11
  Interventions: Behavioral: Online survey
- Middle stage HDGECs: CAG length ≥ 40; DCL = 4, 7 ≤ TFC ≤ 10
  Interventions: Behavioral: Online survey
- Late stage HDGECs: CAG length ≥ 40; DCL = 4, 0 ≤ TFC ≤ 6
  Interventions: Behavioral: Online survey
- Companions of early stage HDGECs
  Interventions: Behavioral: Online survey
- Companions of middle stage HDGECs
  Interventions: Behavioral: Online survey
- Companions of late stage HDGECs
  Interventions: Behavioral: Online survey

INTERVENTIONS:
Behavioral: Online survey — Online survey to capture indirect and out of pocket costs of Huntington's Disease in HDGECs and companions

SUMMARY:
Huntington's disease (HD) is a rare, inherited and progressive neurodegenerative disorder for which hallmark symptoms include movement disorders, loss of cognitive faculties and psychiatric disturbances. With the progression of the disease, patients require increasing level of medical care, caregiver support, and long-term care, which lead to substantial burden of illness. Very little data are available on the direct or indirect costs for HD. The direct medical costs of HD in the US have been summarized from retrospective commercial and Medicaid claims data analysis. The indirect and out-of-pocket costs of HD in the US have not been quantified. This study will help to bridge these gaps.

This study is a single-assessment, cross-sectional online survey administered to Huntington disease gene expansion carriers (HDGECs) and companions of HDGECs by HD stage to understand the indirect and out-of-pocket costs of Huntington's disease in the US.

DETAILED DESCRIPTION:
The survey collects the following data from each HDGEC and companion:

1. Participant demographics (for HDGECs and companion)
2. Informal care received (for HDGECs only)
3. Out of pocket HD costs (for HDGECs and companion)
4. Current employment status (for HDGECs and companion)
5. Non-work and work care giving time that companion spends taking care of HDGEC (for companion only)
6. Work Productivity and Activity Impairment (WPAI) Questionnaire (for HDGECs and companion)

ELIGIBILITY:
Inclusion Criteria for HDGECs:

* Identified as an active participant in Enroll-HD (participants who have completed their last on site Enroll-HD visit within approximately 15 months)
* Able to provide online or written informed consent. A LAR for HDGEC can provide written consent, if applicable
* Identified as a participant with clinically diagnosed HD and has a CAG length ≥ 40
* Site PI has access to HDGEC's medical records for the purpose of completing the Resource Utilization Questionnaire
* Able to speak and understand both verbal and written English
* Has adult onset of disease (disease symptoms manifested at age 20 years or older)
* Has access to a computer/tablet/smartphone (if compatible) and internet services

Stage classification of HDGECs:

1. Early stage HDGEC: CAG length ≥ 40; DCL = 4, TFC ≥ 11
2. Middle stage HDGEC: CAG length ≥ 40; DCL = 4, 7 ≤ TFC ≤ 10
3. Late stage HDGEC: CAG length ≥ 40; DCL = 4, 0 ≤ TFC ≤ 6

Exclusion Criteria for HDGECs:

HDGECs will be excluded from the study if they have significant cognitive or any other impairment sufficient to interfere with study associated tasks as judged by the Site PI or Site PI's designee (exceptions will be made if a companion/LAR completes the survey on their behalf).

Inclusion criteria for companions:

* Able to provide online or written informed consent
* Identified as the primary provider (unpaid) of supportive care of an HDGEC (HDGEC must be an Enroll-HD participant and have a CAG length ≥ 40 and have adult onset of disease (disease symptoms manifested at age 20 years or older))
* Able to speak and understand both verbal and written English
* Aged 21 years or older at time of survey
* Has access to a computer/tablet/smartphone (if compatible) and internet services and has the technical skills required to complete an online survey

Exclusion Criteria for companions:

Companions will be excluded from the study if they are identified as paid or salaried caregivers; however, the HDGECs for whom they care may still be included in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HDGECs: Participant in Enroll-HD with clinically diagnosed HD and a cytosine, adenine, guanine (CAG) length ≥ 40, who meets the protocol inclusion criteria and none of the exclusion criteria.
  Companions: Primary provider (unpaid) of supportive care for an HDGEC (this HDGEC must be an active participant of Enroll-HD Study, have a CAG ≥ 40, have an adult onset of disease (disease symptoms manifested at age 20 years or older), and a DCL=4)), who meets the protocol's companion inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2020-06-21 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Quantify the indirect costs associated with productivity loss for HDGECs and companions | 12 months
  Productivity loss is measured by annual lost wages and it is collected in the survey's employment questionnaires and WPAI
Quantify out-of-pocket expenses for HDGECs and companions | 12 months
  The indirect costs associated with the total annual out-of-pocket expenses.
Identify the indirect costs associated with informal care received for HDGECs | 12 months
  The total informal care time received during a typical week
Quantify the indirect costs associated with non-work caregiving time for companions | 12 months
  The indirect costs associated with the annual opportunity costs of companion

SECONDARY OUTCOMES:
Identify the reasons for HDGEC and companion's unemployment or underemployment | 12 months
The proportion of Dual Role Companions, differentiated by HD stage of the companion | 12 months
To understand traditional disease staging system based on total functional capacity (TFC) | 12 months
  For HDGECs and Companions: Understand how the traditional disease staging system, based on the TFC score, relates to a staging system based on resource utilization questionnaire and comorbid conditions developed in Divino et al. (2013)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Rocky Mountain Movement Disorder, P.C., Englewood, Colorado
  - University of South Florida, Tampa, Florida
  - Hereditary Neurological Disease Centre, Inc., Wichita, Kansas
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided